CLINICAL TRIAL: NCT01392833
Title: Steroids and Azathioprine in Early and Advanced IgA Nephropathy: Amendments to a Prospective Randomised Multicenter Trial
Brief Title: Steroids and Azathioprine in Advanced IgAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A. Manzoni Hospital (Other)
Responsible Party: Claudio Pozzi, Ospedale E. Bassini and A. manzoni Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IgAzaIRC
Record Dates: First submitted 2011-07-05; First posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-03

CONDITIONS: IgA Nephropathy; Chronic Kidney Disease
Keywords: iga nephropathy; chronic kidney disease; proteinuria; steroids; azathioprine
MeSH Terms: conditions — Glomerulonephritis, IGA; Renal Insufficiency, Chronic; Proteinuria | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Azathioprine; Adenosine Triphosphate; Prednisone; deltacortene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- steroids (Active Comparator): intravenous methylprednisolone 1 g for three consecutive days at the beginning of months 1, 3 and 5, and oral prednisone 0.5 mg/kg every other day for six months followed by oral prednisone 0.2 mg/kg every other day for a further six months.
  Interventions: Drug: methylprednisolone; Drug: prednisone
- steroids plus azathioprine (Experimental): intravenous methylprednisolone 1 g for three consecutive days at the beginning of months 1, 3 and 5, and oral prednisone 0.5 mg/kg every other day plus azathioprine 1.5 mg/kg/day for six months followed by oral prednisone 0.2 mg/kg every other day plus azathioprine 50 mg/day for a further six months.
  Interventions: Drug: methylprednisolone; Drug: azathioprine; Drug: prednisone

INTERVENTIONS:
Drug: methylprednisolone — intravenous methylprednisolone 1 g for three consecutive days at the beginning of months 1, 3 and 5
  Other Names: solumedrol
Drug: azathioprine — azathioprine 1.5 mg/kg/day for six months followed by azathioprine 50 mg/day for a further six months.
  Other Names: azatioprina
  Arms: steroids plus azathioprine
Drug: prednisone — prednisone 0.5 mg/kg every other day followed by prednisone 0.2 mg/kg every other day for a further six months.
  Other Names: deltacortene

SUMMARY:
Some years ago the investigators designed a randomised trial to prospectively evaluate whether adding low-dose azathioprine (1.5 mg/kg/day for six months) to steroids (methylprednisolone 1 g i.v. for three consecutive days at months 1, 3 and 5, plus oral prednisone 0.5 mg/kg every other day for six months) can improve long-term renal survival in adult IgAN patients with proteinuria higher than 1g/24 hours and plasma creatinine <=2.0 mg/dl.

In order to test the efficacy of the combination of steroids with azathioprine at various degree of renal function deterioration by extending the trial to patients with more advanced disease (serum creatinine higher or equal to 2 mg/dl) without any time limit for renal biopsy. Treatment will last one year: methylprednisolone 1 g i.v. for three consecutive days at the beginning of months 1, 3 and 5, followed by oral prednisone 0.5 mg/kg every other day for six months, then 0.2 mg/kg every other day for further 6 months. The primary outcome was renal survival (a 50% increase in plasma creatinine from baseline); the secondary outcomes were proteinuria over time and the number and types of adverse events in the two groups assessed every month for the first six months, every two months from the 6th to the 12th month and every three months thereafter. The planned duration of follow up is five years.

DETAILED DESCRIPTION:
It is know well established that IgAN outcome is often unfavourable, with end-stage renal disease (ESRD) occurring in 5-25% of cases within ten years and in 25-50% of cases within 20 years. The degree of impairment in renal function at presentation is certainly an important predictor of this poor outcome. However, although high serum creatinine at the time of diagnosis may allow the detection of patients who are more likely to progress (and perhaps may get some benefit from therapy), no established treatment exists in advanced IgAN. This is likely explained by the fact that renal impairment is often associated with renal biopsy indexes of chronicity such as glomerular sclerosis, tubulointerstitial atrophy or fibrosis. It has also been suggested that in this disease, as in other chronic nephropathy, there is "a point of no return" after which non-immunological mechanisms have been considered to play a central role in a relentless progression.

Most patients with IgAN develop ESRD in middle age and this represents not only a significant problem for the patient itself but also a social and economic burden for society as a whole. For this reason, while waiting for more specific therapies able to complete prevent progression in IgAN, the possibility of delaying the beginning of renal replacement therapy of some years could be considered an important goal in these patients.

In this regard, the investigators were impressed from the results of an uncontrolled retrospective study of combined treatment with corticosteroids for 18 months and azathioprine for 24 months. Although the treatment seemed to be ineffective in the patients with normal renal function (because of the very low number of events in this very-slowly progressive group) and the lack of randomisation led to a severe bias concerning the choice of the patients to be treated (higher risk patients), in those with impaired renal function, a smaller percentage of treated subjects had a progressive course (20.5% vs 63.4%, p < 0.001). Similarly, Tsuruya et al. retrospectively found that combination therapy with prednisolone and cyclophosphamide was effective in reducing urinary protein excretion and in slowing the rate of progression in histologically advanced IgAN.

Given all these consideration, the investigators decided to test the efficacy of the combination of steroids with azathioprine at various degree of renal function deterioration by extending the trial to patients with more advanced disease (serum creatinine > 2 mg/dl). Considering the high likelihood of these patients to have a certain degree of sclerosis and that in focal segmental glomerulosclerosis longer treatments seem to lead to slightly better results in term of achievement and maintenance of partial and complete remissions, in the patients of amendment II the investigators decided to continue the treatment with steroids and azathioprine at a very low dose for other six months, with an overall one-year treatment duration.

Study design The patients are randomly allocated to treatment with steroids (methylprednisolone 1 g i.v. for three consecutive days at the beginning of months 1, 3 and 5, plus oral prednisone 0.5 mg/kg every other day for six months, then 0.2 mg/kg every other day for other six months) plus azathioprine 1.5 mg/kg/day for six months and 50 mg/day for other six months (experimental group) or steroids alone (methylprednisolone 1 g i.v. for three consecutive days at the beginning of months 1, 3 and 5, plus oral prednisone 0.5 mg/kg every other day for six months, then 0.2 mg/kg every other day for other six months) (control group).

If leukocyte count is between 3,000 and 5,000 mmc the dose of azathioprine will be halved; if leukocyte count is below 3,000 mmc, azathioprine will be suspended.

The planned duration of follow up is five years. Similarly to the original protocol, in the presence of proteinuria relapses without an increase in plasma creatinine of more than 50% from baseline, patients of both amendments who have experienced complete or partial remission of proteinuria may be treated again with the same schedule (not before six months after the end of the previous treatment).

All patients will be administered diuretics, antihypertensive drugs and antiplatelet agents as needed. Cyclosporin, immunosuppressive drugs other than azathioprine and anti-inflammatory drugs will not be allowed. ACE-inhibitors and angiotensin II receptor antagonists will be allowed for the treatment of hypertension. Given the importance of blood pressure control in slowing down chronic renal failure progression, a target blood pressure of 130/80 mmHg is warranted.

Treatment allocation Similarly to the original protocol, patients will be randomly allocated to one of the two treatment groups (steroids alone or steroids plus azathioprine). A 48-month recruitment period is estimated.

Trial procedures Patients considered eligible on the basis of the inclusion/exclusion criteria are provided with information concerning the study and asked their informed consent.

Patients will be examined at baseline, and every month for the first six months, every two months from the 6th to the 12th month and every three months thereafter. At each visit, the patients will be asked about their clinical symptoms, possible treatment complications and drug consumption. Their body weight, blood pressure, plasma creatinine levels, hemocrome with leukocyte and platelet counts, total plasma proteins, serum glucose, AST, ALT, GGT, bilirubin, alkaline phosphatase, 24-hour urinary protein excretion will be also measured and recorded.

Histological evaluation Given that renal biopsy is not required to be recent, histological lesions could not reflect the actual state of the disease at the time of randomisation. For this reason, the histological evaluation will not be performed in the patients.

Statistical analysis The results of the trial will be evaluated by intention-to-treat analysis. The primary endpoint will be the progression of renal disease, estimated on the basis of 50% increase of baseline plasma creatinine levels. The doubling of plasma creatinine from baseline will also be considered as a primary end-point. Secondary end-points will be the evolution of proteinuria over time (complete or partial remission respectively defined as proteinuria < 0.2 g/24h and the halving of baseline proteinuria), the number of relapses (defined as proteinuria equal or higher than baseline) and the number and types of adverse events in the two groups assessed every month for the first six months, every two months from the 6th to the 12th month and every three months thereafter. Renal survival without an endpoint will be analysed by means of the Kaplan-Meier method and the two groups will be compared using the log-rank and Breslow tests. Multivariate analysis based on Cox's regression proportional hazards model will be used to estimate the relative risk associated with possible prognostic factors such as sex, age, plasma creatinine levels, proteinuria, arterial hypertension, macroscopic hematuria, ACE-inhibitors, angiotensin II receptor antagonists.

The minimum length of the follow up will be of five years.

ELIGIBILITY:
Inclusion Criteria:

* Serum creatinine higher or equal to 2.0 mg/dl
* Proteinuria higher or equal to 1g/24g for at least three months
* No time limits for renal biopsy

Exclusion Criteria:

* Steroids and/or cytotoxic drugs (used for more than three months) in the previous three years
* Contraindications to steroids or azathioprine
* Diabetes
* Severe hypertension (diastolic blood pressure > 120 mmHg)
* Liver disease
* Infections
* Active peptic-ulcer disease
* Malignancies
* Pregnancy
* Secondary IgAN

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 1999-12; Primary Completion 2006-11 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
renal survival | five years
  time to a 50% increase in serum creatinine from baseline

SECONDARY OUTCOMES:
proteinuria | at six month and during follow up
  proteinuria changes
adverese events (possible treatment related) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: claudio pozzi, md, Principal Investigator — A. Manzoni Hospital, ospedale G. bassini